CLINICAL TRIAL: NCT05543226
Title: The Effect of PHGG-rich Enteral Nutrition to on the Infection in Liver Transplant Recipients: A Prospective, Double-blind, Randomized Controlled Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-KY-029
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-03

CONDITIONS: Infections
MeSH Terms: conditions — Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PHGG (Experimental)
  Interventions: Drug: PHGG-rich enteral nutrtiion
- without PHGG (Placebo Comparator)
  Interventions: Drug: PHGG-rich enteral nutrtiion

INTERVENTIONS:
Drug: PHGG-rich enteral nutrtiion — PHGG-rich enteral nutrition

SUMMARY:
To known the effect of PHGG-rich enteral nutrition to on the infection in liver transplant recipients

ELIGIBILITY:
Inclusion Criteria:

1. liver transplant recipients
2. age from 18 to 80 years old
3. APACHE II score >12
4. There is an indication for enteral nutrition and it is expected to require oral or tube feeding for more than 7 days
5. there is no intra-abdominal infection or bloodstream infection

Exclusion Criteria:

1. Severe cardiac, kidney and lung dysfunction
2. bowel obstruction, intestinal perforation, intestinal leakage before operation
3. Roux and Y anastomosis during liver transplant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of infections after liver transplantation | 30 days
  the incidence of infections after 30 days of the liver transplantation

IPD SHARING:
Plan to Share IPD: No